CLINICAL TRIAL: NCT03989505
Title: Proenkephalin ANd Creatinine in the Prediction of Cardiac Contrast-Associated Kidney Events
Brief Title: Proenkephalin for Prediction of Contrast-Associated Kidney Events
Acronym: PANCAKE
Status: Completed | Type: Observational
Sponsor: Dr. med. Mahir Karakas (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Mahir Karakas, Coordinating Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: PANCAKE
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Contrast-induced Nephropathy; Acute Kidney Injury; Coronary Artery Disease
Keywords: CIN; Coronary Angiography; Contrast; Angiography
MeSH Terms: conditions — Acute Kidney Injury; Coronary Artery Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A venous blood sample (10 ml EDTA, 10ml Serum) for storage and further analysis
  * A venous blood sample (Buffy Coat) for DNA Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: 214 consecutive patients undergoing contrast-enhanced diagnostic and/ or therapeutical intervention in the cath lab of the University Heart Center Hamburg
  Interventions: Diagnostic Test: blood-draw for biomarker analyses

INTERVENTIONS:
Diagnostic Test: blood-draw for biomarker analyses — Blood will be drawn at three time-points: immediately before catherization, 12-24 hours after catheterization and 4-8 weeks after discharge. Creatinine will be measured for endpoint definition, while the markers urea, CRP (C-reactive protein), NGAL (neutrophil gelatinase-associated lipocalin), KIM-1 (kidney injury marker-1), cystatin C, suPAR (soluble urokinase-type plasminogen activator receptor), and penKid will be measured as biomarkers of interest.

SUMMARY:
Currently, contrast-induced kidney injury cannot be diagnosed on the day of cardiac catheterization. Recently, proenkephalin (penKid) was introduced as a new glomerular filtration marker. The aim of this study is to investigate whether the change in penKid level allows for early detection of affected patients.

DETAILED DESCRIPTION:
Use of contrast media is necessary for diagnostic imaging and percutaneous coronary intervention. However, contrast-induced kidney injury, a complication of contrast use, has been identified as the most frequent cause of hospital-acquired acute kidney injury and is associated with poor prognosis. Currently, contrast-induced kidney injury cannot be diagnosed on the day of cardiac catheterization or on the following day, when the majority of patients who undergo elective cardiac catheterization are discharged from the hospital in the real-world setting. Recently, proenkephalin (penKid) was introduced as a new glomerular filtration marker, which is capable of identifying normal subjects at high risk of future decline in renal function. The aim of this study is to investigate whether the change in penKid level on the day following cardiac catheterization can predict kidney injury before hospital discharge and thus allows for early detection of affected patients.

For this purpose a total of 214 consecutive patients who undergo routine cardiac catherization will be recruited, and blood will be drawn at three time-points: immediately before catherization, 12-24 hours after catheterization and 4-8 weeks after discharge. Creatinine will be measured for endpoint definition, while the markers urea, CRP (C-reactive protein), NGAL (neutrophil gelatinase-associated lipocalin), KIM-1 (kidney injury marker-1), cystatin C, suPAR (soluble urokinase-type plasminogen activator receptor), and penKid will be measured as biomarkers of interest. The main outcome measure is sustained kidney injury (SKI), which is defined as an increase above 20% in serum creatinine between time-points 1 and 3. The main test is whether the change in biomarkers between baseline and immediately before discharge (time-points 1 and 2) can predict the development of sustained kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Planned elective or urgent coronary or non-coronary angiography with iodinated contrast media
* Ability to provide informed consent

Exclusion Criteria:

* Current use of renal replacement therapy/hemodialysis
* life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing coronary or non-coronary angiography with iodinated contrast media at the University Heart Center Hamburg
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sustained kidney injury | Time period between the two time-points: immediately before catherization and 4-8 weeks after discharge
  defined as an increase above 20% in serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, Principal Investigator — University Heart Center Hamburg; Johannes F Geng, MD, Principal Investigator — University Heart Center Hamburg
Locations (1):
- University Heart Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided